CLINICAL TRIAL: NCT04526834
Title: Phase 1 Study of CD30-Directed Genetically Modified Autologous T-Cells (CD30.CAR-T) in Patients With Relapsed or Refractory CD30 Positive Non-Hodgkin Lymphoma
Brief Title: Phase 1 Study of Autologous CD30.CAR-T in Relapsed or Refractory CD30 Positive Non-Hodgkin Lymphoma
Acronym: CERTAIN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tessa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESSCAR002
Record Dates: First submitted 2020-08-20; First posted 2020-08-26 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Anaplastic Large Cell Lymphoma; Peripheral T Cell Lymphoma; Extranodal NK/T-cell Lymphoma; Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B-Cell Lymphoma (PMBCL)
Keywords: CD30, r/r NHL, DLBCL, ALCL, ENKTCL, PMBCL, PTCL, adult
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Peripheral; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD30 positive NHL subtypes (Experimental): (ALCL, PTCL-NOS, ENKTCL, DLBCL-NOS, PMBCL)
  Dose Level 1
  Dose Level 2
  Dose Level 3
  Interventions: Drug: CD30.CAR-T

INTERVENTIONS:
Drug: CD30.CAR-T — Bendamustine and Fludarabine (3 days)
  Dose level 1: 2 x 108 cell/m2 CD30.CAR-T (Day 0)
  Dose level 2: 4 x 108 cell/m2 CD30.CAR-T (Day 0)
  Dose level 3: 6 x 108 cell/m2 CD30.CAR-T (Day 0)
  Other Names: CD30-directed genetically modified autologous T cells

SUMMARY:
This is a phase 1 study to evaluate safety and dose-limiting toxicity of autologous CD30.CAR-T in subjects with relapsed or refractory CD30+ Non-Hodgkin Lymphoma

DETAILED DESCRIPTION:
Adult patients with relapsed or refractory CD30-positive Non-Hodgkin Lymphoma who have failed standard available therapies and who meet eligibility criteria will have blood drawn to manufacture the CD30.CAR-T cells.

CD30.CAR-T cells will be infused once following the completion of lymphodepleting chemotherapy with Bendamustine and Fludarabine.

Subjects will be closely monitored for DLT and safety.

ELIGIBILITY:
Inclusion Criteria:

Eligibility is determined priori to leukapheresis. Patients must satisfy the following criteria to be enrolled in this study:

1. Signed Informed Consent Form
2. Male or female patients who are 18-75 years of age
3. Histologically confirmed ALCL, PTCL- NOS, ENKTCL nasal type, DLBCL-NOS and PMBCL
4. Relapsed or refractory CD30-positive NHL who have failed all available standards of therapy. Patients may or may not have received an autologous or allogeneic HSCT CD30-positive tumor
5. At least 1 measurable lesion according to the Lugano Classification
6. ECOG PS of 0 to 1 or equivalent Karnofsky PS Anticipated life expectancy >12 weeks

Exclusion Criteria:

1. CNS involvement by malignancy
2. Inadequate laboratory abnormalities at screening:

   Hgb ≤ 8.0 g/dL Total bilirubin > 1.5 x ULN (>2 x ULN for patients with Gilbert's syndrome) AST and ALT ≥ 5 x ULN CrCL ≤ 45 mL/min (as measured by Cockcroft-Gault equation) ANC ≤ 1000/uL Platelets ≤75,000/uL PR or INR >1.5 x ULN aPTT> 1.5 x ULN
3. Active uncontrolled bleeding or a known bleeding diathesis
4. Inadequate pulmonary function defined as pulse oximetry < 90% on room air
5. Ongoing treatment with immunosuppressive drugs including calcineurin inhibitions, TNFalpha, mTOR, etc or chronic systemic corticosteroids (>10 mg/day prednisone or equivalent for >48 hours)
6. Received prior therapy of:

   Anti-CD30 Ab based therapy within the previous 8 weeks Previous CD30.CAR-T investigational product Bi-specific CD30 Ab within the previous 8 weeks Allogenic HSCT in the last 180 days Autologous HSCT within 90 days
7. Active GVHD requiring immune suppression regardless of grade
8. HIV positive
9. Active HBV and/or HCV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and dose limiting toxicities (DLT) of autologous CD30.CAR-T and establish the recommended Phase dose | Day 0 to 28 for DLT
  Incidence of DLTs and occurrence of study related adverse events

SECONDARY OUTCOMES:
To evaluate pharmacokinetics of autologous CD30.CAR-T | Start of infusion of CD30.CAR-T (Day 0) until year 5
  AUC (copies/ug DNA over time)
Objective Response Rate (ORR) | Start of CD30.CAR-T (Day 0) until progressive disease or start of new cancer therapy, whichever comes first, up to one year
  ORR
Duration of Response (DOR) | Start of CD30.CAR-T (day 0) until progressive disease or death, whichever comes first, up to one year
  DOR
Progression Free Survival (PFS) | Start of CD30.CAR-T (Day 0) until progressive disease or death, whichever comes first, up to one year
  PFS

CONTACTS AND LOCATIONS:
Overall Officials: Sairah Ahmed, Principal Investigator — MD Anderson
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Centre, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338